CLINICAL TRIAL: NCT07312630
Title: Clinical Study of LV009 Injection for the Treatment of Relapsed/Refractory CD19-Positive Hematologic and Lymphoid Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-012-8
Record Dates: First submitted 2025-09-29; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin Lymphoma (NHL); Acute Lymphoblastic Leukemia (ALL), Adult
Keywords: CD19; CAR-T
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: LV009 Injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection of CD19-Targeted Chimeric Antigen Receptor T Cells (Experimental): A dose escalation was conducted using four fixed doses of LV009 injection solution: 0.3 × 10^9, 0.6 × 10^9, 1.2 × 10^9, and 2.4 × 10^9 TU.
  Interventions: Biological: LV009 Injection Infusion

INTERVENTIONS:
Biological: LV009 Injection Infusion — A dose escalation was conducted using four fixed doses of LV009 injection solution: 0.3 × 10^9, 0.6 × 10^9, 1.2 × 10^9, and 2.4 × 10^9 TU.

SUMMARY:
Evaluate the safety, pharmacokinetic (PK) characteristics, and pharmacodynamic (PD) characteristics of LV009 injection in subjects with relapsed/refractory CD19-positive hematologic malignancies.

DETAILED DESCRIPTION:
Within each dose group, the next subject may be dosed after the previous subject has completed at least 14 days of safety observation. Following the assessment of dose-limiting toxicity (DLT) within 28 days after the last subject in each dose group completed a single dose, and upon approval by the Safety Review Committee (SRC) based on clinical safety data to proceed to the next dose group, enrollment and treatment for the next dose group may commence. If one DLT occurs among the first three subjects in a dose group, three additional subjects must be added to that group (bringing the total to six subjects for DLT assessment): If no DLT occurs in the 3 additional subjects, dose escalation continues. If 1 DLT occurs in the 3 additional subjects, dose escalation is halted. If >1 DLT occurs in the 3 additional subjects, dose escalation is halted, and the dose must be reduced by one level to continue enrolling 3 subjects for DLT assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old (inclusive of both age limits), no gender restrictions, no racial restrictions
* Expected survival time exceeds 12 weeks
* ECOG performance status 0-2
* Meets the NCCN guidelines' criteria for recurrence/refractory disease and is diagnosed with CD19-positive hematologic malignancies, including non-Hodgkin lymphoma (NHL) and acute lymphoblastic leukemia (ALL)
* Liver and kidney function, as well as cardiopulmonary function, meet requirements.
* Absolute lymphocyte count ≥ 0.5 × 10⁹/L; platelet count ≥ 50 × 10⁹/L; CD3-positive T cells ≥ 150 cells/μL.
* Subjects must have a body temperature ≤ 38°C (excluding tumor fever) within 24 hours prior to study drug infusion and must not have significant active infection.
* Within 5 days prior to the study drug infusion, subjects must not receive therapeutic doses of corticosteroids (>5 mg/day of prednisone or other equivalent doses of corticosteroids) or other immunosuppressive agents.

Exclusion Criteria:

* Patients deemed by the investigator to require long-term use of immunosuppressive agents during screening should be excluded.
* Patients who have experienced a cerebrovascular accident or seizure within the six months prior to signing the informed consent form must be excluded.
* Patients with malignant tumors other than the study disease must be excluded (only patients with carcinoma in situ may be considered for inclusion).
* Hepatitis B surface antigen (HBsAg) positive; Hepatitis B core antibody (HBcAb) positive with peripheral blood hepatitis B virus (HBV) DNA titer outside normal reference range; Hepatitis C virus (HCV) antibody positive with peripheral blood hepatitis C virus (HCV) RNA positive; Human Immunodeficiency Virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA positive; Syphilis positive. (Patients meeting any criterion in this section must be excluded.)
* Patients with severe cardiac conditions must be excluded, including but not limited to: unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] class ≥ III), and severe arrhythmias.
* Patients judged by the investigator to have unstable systemic diseases must be excluded, including but not limited to those with severe liver, kidney, or metabolic diseases requiring medication.
* Patients with chronic progressive neurological diseases should be excluded.
* Patients who have not recovered from acute toxic effects following prior treatment must be excluded.
* Patients with active infections requiring systemic treatment or uncontrolled infections should be excluded (patients with mild urogenital tract infections and upper respiratory tract infections may be considered for inclusion).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
TEAE | From the start of infusion of the study drug to 3 months after drug infusion
  According to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
(Tmax) | Within 28 days after the transfusion and within 90 days after the transfusion
  Time to peak concentration of CD19 CAR-T expansion in peripheral blood following administration of LV009 injection
(Cmax) | Within 28 days after the transfusion and within 90 days after the transfusion
  Maximum concentration of CD19 CAR-T expansion in peripheral blood following administration of LV009 injection
AUC | Within 28 days after administration of LV009 injection
  Area under the curve of CD19 CAR-T expansion in peripheral blood 28 days after administration of LV009 injection

CONTACTS AND LOCATIONS:
Locations (1):
- PersonGen.Anke Cellular Therapeutice Co., Ltd., Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
Because the patent rights have not yet been determined.